CLINICAL TRIAL: NCT03881774
Title: Clinical Study of Cord Blood Derived CAR-T Cells in Patients With Refractory/Relapsed B Cell Leukemia/Lymphoma Who Are Failed for Autologous CAR-T Cells or Autologous CAR-T Can Not be Prepared
Brief Title: Cord Blood Derived CAR-T Cells in Refractory/Relapsed B Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Henan Hualong Biotechnology Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH CART 2-4
Record Dates: First submitted 2019-03-16; First posted 2019-03-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Refractory; Relapsed; B Cell Lymphoma; B Cell Leukemia
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Leukemia, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: CAR-T cell group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): cord blood derived CAR T cells group
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — collecting cord blood for CAR-T cells culture; three days later, FC regimen (fludarabine 30mg/m2/d x 3, cyclophosphamide 600-800mg/m2/d x 2) another two days later, transfusing CAR-T cell with a dose of 0.5-3x106/kg
  Other Names: cord blood derived CAR-T cells

SUMMARY:
Evaluation the safety and efficacy of cord blood-derived CAR-T cells in patients with relapsed/refractory B cell leukemia/lymphoma whose disease relapsed after autologous CAR-T cells therapy or who fail to preparation for autologous CAR-T cells

DETAILED DESCRIPTION:
CAR-T cells therapy is the preferred option for relapsed/refractory B cell leukemia/lymphoma. However, some patients will relapse after CAR-T cells therapy, and because of previous multicycles chemotherapy it's very difficult to abtain enough lymphocytes for preparation of antologous CAR-T cells. The exploration of alternative source of lymphocytes for CAR-T cells preparation has important clinical implications for such patients. We evaluated the efficacy and safety of cord blood-derived CAR-T cells in such patients, and to explore effective treatment options for such patients.

ELIGIBILITY:
Inclusion Criteria:

* expected lifespan >3 months
* patients with refractory/relapsed B cell leukemia/lymphoma whose diseases relapse after autologous CAR-T cells or the preparation for autologous CAR-T cells fails
* KPS >70
* for patients with lymphoma, at least one measurable lesion according to RECIST 1.1
* enough function of heart, liver, kidney and bone marrow
* no history of severy allergy
* no other serious diseases that conflict with this plan
* no other history of malignancy
* no serious mental illness
* patients and their families members agree to participate in this clinical study and sign the Informed Consent Form

Exclusion Criteria:

* pregnant or lactating women
* vevere infectious or viral diseases
* active hepatitis B or C viral hepatitis
* Patients who have used large amounts of glucocorticoids or other immunosuppressive agents within the last 4 weeks
* participated in other clinical studies in the past 3 months or who have been treated with other gene products;
* others that other investigators consider not suitable for this clinical study

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
occurrence of study related adverse events | one year
  safety of CAR-T cells

SECONDARY OUTCOMES:
objective response rate | three months
  the proportion of patients with CR or PR
progression-free survival | one year
  from the date of enrollment to the first date of progression detected
overall survival | one year
  from the date of enrollment to the date of death
copy number of CAR-T | six months
  copy number of CAR-T in blood and bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, Dr., Study Chair — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No